CLINICAL TRIAL: NCT03043261
Title: Effective Management of Emotional Response to Generate Well-Being Post-HF Exacerbation
Acronym: EMERGE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Pro00078272
Record Dates: First submitted 2017-02-02; First posted 2017-02-06 (Estimated); Last update posted 2018-05-07 (Actual); Status verified 2018-05

CONDITIONS: Congestive Heart Failure
Keywords: CHF
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Psycho-Behavioral Intervention (Experimental): Williams LifeSkills modules which cover 10 core skills designed to improve coping skills, stress management and interpersonal relationships: 1) being aware of negative thoughts and feelings, 2) making a decision, 3) deflection skills, 4) problem solving or action skills, 5) assertion, 6) saying "no", in addition to the following preventive skills: 7) speaking up, 8) listening, 9) empathy and 10) increasing positives
  Interventions: Behavioral: Williams LifeSkills

INTERVENTIONS:
Behavioral: Williams LifeSkills — Online multi-media interactive training modules which address 10 core skills to improve coping, stress management and interpersonal relationships.

SUMMARY:
EMERGE is a PI-initiated feasibility study that aims to evaluate the accessibility, usability, effectiveness and relevance of an integrated psycho-behavioral intervention on heart failure patients in order to increase support, outreach and general well-being of these patients following hospitalization due to heart failure exacerbation.

ELIGIBILITY:
Inclusion Criteria:

* Adult male and female patients, age ≥ 18 hospitalized at Duke inpatient service because of heart failure
* NYHA Class ≥ II

Exclusion Criteria:

* Significant cognitive impairment, indicated as a mini-mental state exam (MMSE) total score of 23 or lower
* Lack of convenient internet access outside of hospital
* Alcohol or other drug dependence/abuse within past 90 days as evaluated by review of medical record and patient interview (SCID)
* Severe physical disability (visual, sensory or motor) that may interfere with study participation (assessment, online interactive learning)
* History or presence of psychoses, bipolar disorder, and/or severe personality disorders as evaluated by review of medical record and patient interview (SCID)
* Life-threatening co-morbidity with the likelihood of 50% mortality in one year
* Active suicidal ideations
* Female patients of childbearing potential
* Treatment with electroconvulsive therapy or transcranial magnetic stimulation within past 90 days
* Uncorrected hypothyroidism or hyperthyroidism

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2018-01-29 (Actual); Primary Completion 2018-04-07 (Actual); Study Completion 2018-04-07 (Actual)

PRIMARY OUTCOMES:
Subject retention | 6 month
  Percentage of subjects who complete the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Wei Jiang, M.D., Principal Investigator — Duke University
Locations (1):
- Pamela Bonner, Durham, North Carolina, United States